CLINICAL TRIAL: NCT04176471
Title: The TIME STUDY: A Randomized Controlled Trial of Therapeutic Hypothermia for Infants With Mild Encephalopathy in California
Brief Title: TIME Study: Therapeutic Hypothermia for Infants With Mild Encephalopathy
Acronym: TIME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stanford University (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Sonia Bonifacio, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 53274
Record Dates: First submitted 2019-11-14; First posted 2019-11-25 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Hypoxic-Ischemic Encephalopathy Mild; Neonatal Encephalopathy
MeSH Terms: interventions — Hypothermia, Induced

STUDY DESIGN:
Intervention Model Description: A total of 68 neonates with mild HIE will be enrolled and randomized to therapeutic hypothermia (33.5°C ± 0.5°C for 72 hours plus 6 hours of rewarming) or normothermia (36.5-37.3°C for 72 hours ) with targeted temperature management. Each treatment group will have 34 patients. Participants randomized to normothermia who develop signs of moderate-severe HIE in the first 24 hours after birth will be crossed over to the treatment arm, as therapeutic hypothermia is the standard of care treatment for neonates with moderate-severe HIE.
Who Masked: Outcomes Assessor
Masking Description: Assessors of neurodevelopmental outcome at 12-14 months of age will be blinded to the allotted treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Hypothermia (Experimental): Therapeutic hypothermia will be achieved using a servo-controlled temperature regulating blanket that is approved for use in neonates and is currently used for the treatment of neonates with moderate-severe HIE. The goal target temperature is 33.5°C ± 0.5°C for 72 hours and the subject will then be rewarmed at a rate of 0.5°C per hour to a goal of 36.5°C.
  Interventions: Other: Therapeutic Hypothermia
- Normothermia (Active Comparator): Normothermia will be achieved using a servo-controlled temperature regulating blanket with the temperature goal of 36.5-37.3°C for 72 hours.
  Interventions: Other: Normothermia

INTERVENTIONS:
Other: Therapeutic Hypothermia — Therapeutic hypothermia involves use of a servo-controlled device and blanket to lower the core body temperature by 3°C for 72 hours followed by a period of re-warming in which the temperature is increased by 0.5°C per hour for 6 hours until normothermia is achieved.
  Arms: Therapeutic Hypothermia
Other: Normothermia — Normothermia will be achieved using the same servo-controlled device and blanket to assure normothermia of the control arm. The goal temperature for normothermia is 36.5-37.3°C for 72 hours.
  Arms: Normothermia

SUMMARY:
The TIME study is a randomized, controlled trial to evaluate impact on early measures of neurodevelopment and the safety profile of therapeutic hypothermia in term neonates with Mild Hypoxic-Ischemic Encephalopathy who are < 6 hours of age. Neurodevelopmental outcome will be assessed at 12-14 months of age. The study will enroll 68 neonates randomized to therapeutic hypothermia or normothermia across 5 centers in California.

DETAILED DESCRIPTION:
The TIME study is a multi-center randomized, controlled trial of Therapeutic Hypothermia (TH) (33.5°C ± 0.5° for 72 hours) versus normothermia using targeted temperature management, initiated within 6 hours after birth in term neonates with Mild Hypoxic-Ischemic Encephalopathy (HIE). Mild encephalopathy will be identified using the 6 component modified Sarnat exam as in the Neonatal Research Network of the National Institute of Child Health and Human Development trials of TH for moderate-severe encephalopathy and will be expanded to include features of mild encephalopathy. Eligible subjects must demonstrate ≥ 2 exam abnormalities (mild, moderate, severe) but without evidence of moderate-severe encephalopathy (≥ 3 moderate or severe features). The primary outcome is neurodevelopmental outcome at 12-14 months of age. Secondary outcomes include evaluating the safety profile of therapeutic hypothermia in patients with Mild HIE. Therapeutic hypothermia is well tolerated and did not demonstrate serious safety concerns when evaluated in multiple large studies of neonates with moderate-severe HIE. It is now being applied by some practitioners to neonates with Mild HIE without systematic evidence of benefit or potential harm. This data will be necessary in order to develop and larger trial of efficacy to be determined at 2 years of age.

ELIGIBILITY:
Inclusion Criteria (must meet all 3):

1. Neonates born at ≥ 36 0/7 weeks
2. Neonatal signs or contributing factors consistent with an acute peri-partum or intra-partum event (must meet a or b):

   1. pH ≤ 7.0 or Base deficit ≥ 16 in any umbilical cord or baby specimen at ≤ 1 hr of age OR
   2. No umbilical cord or baby blood gas at ≤ 1 hr of age OR pH 7.01-7.15 or Base deficit 10-15.9 in any cord or baby specimen at ≤ 1 hr of age AND at least one of the following

      * Apgar score at 10 min ≤ 5
      * Continued need for resuscitation at 10 min (chest compressions, bag mask ventilation, intubation with positive pressure ventilation)
      * Acute Perinatal Event: uterine rupture, placental abruption, cord accident (prolapse, rupture, knot or tight nuchal cord), maternal trauma, maternal hemorrhage or cardiorespiratory arrest, fetal exsanguination from either vasa previa or feto-maternal hemorrhage
      * Fetal heart rate monitor pattern consistent with acute peripartum or intrapartum event (category III trace: no heart rate variability, presence of recurrent late or variable decelerations, bradycardia, or sinusoidal pattern)
3. Evidence of Mild Encephalopathy on Modified Sarnat Exam.

   * Presence of at least 2 signs of mild, moderate or severe encephalopathy with no more than 2 moderate or severe findings in the 6 tested categories (level of consciousness, spontaneous activity, posture, tone, neonatal reflexes (suck and moro), and autonomic nervous system

Exclusion Criteria:

* Patients < 36 0/7 weeks birthweight < 1800gm; congenital or chromosomal anomaly associated with abnormal neurodevelopment or death; patients with moderate or severe HIE (by Sarnat exam or presence of clinical or electrographic seizures) identified within 6 hours after birth; core body temperature < 34°C for more than 1 hour prior to randomization.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Warner Initial Developmental Evaluation of Adaptive and Functional Skills (WIDEA-FS) | Assessment takes up to 15 minutes and will be conducted at 12-14 months of age
  Warner Initial Developmental Evaluation of Adaptive and Functional Skills (WIDEA-FS) will be assessed at 12-14 months of age. The mean score for a 12 month old normally developing infant is 109 with a standard deviation of 16.5. Higher scores are associated with normal development.
Alberta Infant Motors Scale (AIMS) | Assessment takes up to 15 minutes and will be conducted at 12-14 months of age
  Alberta Infant Motors Scale (AIMS) will be assessed at 12-14 months of age. The AIMS score is determined by assessment of 4 positions and scoring the least and most mature position identified. The score is converted to a percentile for age with those in the 5th to 25th percentile identified as suspicious motor development and those with a score corresponding to < 5th percentile being identified as abnormal motor development.

SECONDARY OUTCOMES:
Percentage of participants with sinus bradycardia | 72 hours
  Investigators will determine the proportion of treated and control subjects who develop sinus bradycardia (HR < 80) during the intervention period (72 hours).
Percentage of participants thrombocytopenia | 72 hours
  Investigators will determine the proportion of treated and control subjects who develop thrombocytopenia (platelet count of < 150 x 109/L) during the intervention period
Percentage of patients who require intubation and mechanical ventilation | 72 hours
  Investigators will determine the proportion of treated and control subjects who require intubation and mechanical ventilation
Percentage of patients with need for central line | 72 hours
  Investigators will determine the proportion of treated and control subjects who have a central line (umbilical or PICC)
Percentage of participants with Persistent Pulmonary Hypertension (PPHN) | 72 hours
  Investigators will determine the proportion of treated and control subjects who have a clinical diagnosis of PPHN or who receive inhaled nitric oxide
Percentage of participants exposed to sedating or analgesic medications | 72 hours
  Investigators will determine the proportion of treated and control subjects who receive narcotics or benzodiazepines
Percentage of participants exposed to inotropic agents | 76 hours
  Investigators will determine the proportion of treated and control subjects who receive inotropic support
Percentage of participants diagnosed with seizures | During initial hospital stay up to 30 days
  Investigators will determine the proportion of treated and control subjects who develop clinical and or electrographic seizures
Age at initiation of feeds | During initial hospital stay up to 30 days from date of admission
  Investigators will determine the age at which enteral feeds are initiated in treated and control patients
Age at full enteral feeds | During initial hospital stay and up to 30 days from date of admission
  Investigators will determine the age at which full enteral feeds or breastfeeding ad lib is achieved in treated and control patients
Percentage of participants who require feeding assistance at discharge | At time of discharge from hospital, up to 30 days from admission
  Investigators will determine the proportion of treated and control patients who require feeding support at discharge (NG tube or G-Tube feeds)
Percentage of participants with fat necrosis and hypercalcemia | From study entry to day of hospital discharge, up to 30 days from admission
  Investigators will determine the proportion of treated and control patients who have a diagnosis of fat necrosis and hypercalcemia
Percentage of participants discharged on anti-convulsant medications | At time of discharge from hospital, up to 30 days from admission
  Investigators will determine the proportion of treated and control patients who are discharged home on anti-convulsant medications
Count of participants with brain injury on MRI | At time of discharge from hospital, up to 30 days from admission
  Investigators will determine the number of treated and control patients who have brain injury on MRI
Length of Hospital Stay | At time of discharge from hospital, up to 30 days from admission
  Investigators will determine the length of hospital stay for treated and control patients
Percentage of participants breastfeeding at discharge | At time of discharge from hospital, up to 30 days from admission
  Investigators will determine the proportion of treated and control patients who are breastfeeding at discharge
Percentage of participants with death and/or hospice at discharge | At time of discharge from hospital, up to 30 days from admission
  Investigators will determine the proportion of treated and control patients who die or are discharged home on hospice

OTHER OUTCOMES:
Age at Randomization | First 24 hours of life
  Age in hours and minutes after birth at randomization
Age at Initiation of Treatment | First 24 hours of life
  Age in hours and minutes after birth at which normothermia or therapeutic hypothermia are initiated
Percentage of participants with disability at 2 years of age | 2 years
  Most enrolled neonates will be followed in high-risk infant follow-up clinics. We will track developmental outcome at 2 years of age for all enrolled patients and determine the proportion of treated and control patients who abnormal measures of neurodevelopment

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Bonifacio, MD, Principal Investigator — Stanford University
Locations (5):
- United States (5):
  - Loma Linda Children's Hospital, Loma Linda, California
  - Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital Orange County, Orange, California
  - Stanford University, Palo Alto, California
  - Rady Children's Hospital, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akula VP, Sriram A, Xu S, Walsh E, Van Meurs K, Cranshaw M, Kuzniewicz MW. Adverse short- and long-term outcomes among infants with mild neonatal encephalopathy. Pediatr Res. 2023 Sep;94(3):1003-1010. doi: 10.1038/s41390-022-02249-8. Epub 2022 Aug 23. PMID 35999380
- [Derived] Blecharczyk E, Lee L, Birnie K, Gupta A, Davis A, Van Meurs K, Bonifacio S, Frymoyer A. Standardized Evaluation of Cord Gases in Neonates at Risk for Hypoxic Ischemic Encephalopathy. Hosp Pediatr. 2022 Jan 1;12(1):29-37. doi: 10.1542/hpeds.2021-006135. PMID 34854918